CLINICAL TRIAL: NCT03219619
Title: Effect of Cap-assisted Esophagogastroduodenoscopy on Observation of Major Duodenal Papilla: a Randomized Non-inferiority Trial
Brief Title: Effect of Cap-assisted Esophagogastroduodenoscopy on Observation of Major Duodenal Papilla
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Yanglin Pan, Associate Professor, Air Force Military Medical University, China
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: KY20170517-3
Record Dates: First submitted 2017-07-13; First posted 2017-07-17 (Actual); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Observation of Major Duodenal Papilla (MDP)

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cap group: Cap-EGD (Experimental): Undergoing cap-assisted esophagogastroduodenoscopy
  Interventions: Device: Cap-EGD
- Duo group: Duo (Active Comparator): Undergoing side-viewing duodenoscope
  Interventions: Device: Duo

INTERVENTIONS:
Device: Cap-EGD — Undergoing cap-assisted endoscopy
  Arms: Cap group: Cap-EGD
Device: Duo — Undergoing side-viewing duodenoscope
  Arms: Duo group: Duo

SUMMARY:
Examination of major duodenal papilla (MDP) using a side-viewing duodenoscope is a golden standard. However, side-viewing duodenoscope is not available in some endoscopic centers. Cap-assisted esophagogastroduodenoscopy (Ca-EGD) using a transparent cap fitted to the tip of the scope has emerged as an alternative method for the observation of MDP. A recent study showed that complete examination of MDP could be achieved in 97% of patients. The investigators hypothesize that Ca-EGD is non-inferior to duodenoscope for the observation of MDP.

DETAILED DESCRIPTION:
Interim analyses were planned to be performed by the data and safety monitoring board after data collection has been completed for 50% of the enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years and < 70 years
* Patients with native MDP who underwent ERCP

Exclusion Criteria:

* Prior surgery in upper GI tract
* Prior history of endoscopic sphincterotomy
* Prior history of MDP treatment
* Known or suspected obstruction of upper GI tract
* Patients in poor condition who may not be suitable for Ca-EGD or duodenoscope
* Pregnancy or lactic women
* Inability to give informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2018-07-20 (Actual); Primary Completion 2018-07-20 (Actual); Study Completion 2018-07-20 (Actual)

PRIMARY OUTCOMES:
Rate of complete examination of MDP | 5 minutes after intubation of the esophagus
  Complete examination is defined by visualization of both proximal and distal ends with orifice of papilla

SECONDARY OUTCOMES:
Endoscopic findings in descending duodenum | 5 minutes after intubation of the esophagus
  All pathological findings which are seen in descending duodenum should be reported (e.g. ampullary adenoma, peripapillary diverticulum, ampullary carcinoma, inflammatory change of papilla, etc)
Overall endoscopic findings | 5 minutes after intubation of the esophagus
  All pathological findings which are seen during the examination should be reported (e.g. reflux esophagitis, gastric cancer, gastric ulcer, duodenal ulcer, etc)
MDP examination time | 5 minutes after intubation of the esophagus
  The times taken for the examination of the MDP (after passing the pylorus until examination of MDP)
MDP examination score | 5 minutes after intubation of the esophagus
  Score 3 when proximal end, distal end and orifice were visualized; Score 2 when either proximal or distal end with orifice were visualized; Score 1 when either proximal or distal end without orifice was visualized; Score 0 when the MDP could not be localized

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Endoscopic center, Xijing Hospital of Digestive Diseases, Xi'an, Shaanxi
  - Department of gastroenterology, Second Affiliated Hospital of Chongqing Medical University, Chongqing

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shi X, Luo H, Ning B, Wang X, Tao Q, Liang S, Zhang R, Chen J, Luo B, Yao S, Pan Y, Guo X, Fan D. Effect of cap-assisted esophagogastroduodenoscopy on examination of the major duodenal papilla: a noninferior, randomized controlled trial. Endoscopy. 2019 May;51(5):427-435. doi: 10.1055/a-0767-6529. Epub 2019 Jan 8. PMID 30620948